CLINICAL TRIAL: NCT04111328
Title: the Effect of Different Drugs and Infusion Ways on Degree of Comfort for Patients Undergoing Spinal Neoplasm Surgery
Brief Title: the Effect of Different Drugs and Infusion Ways on Degree of Postoperative Comfort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jun Wang (Other)
Responsible Party: Sponsor-Investigator, Jun Wang, Professor, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-191-2
Record Dates: First submitted 2019-09-25; First posted 2019-10-01 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-07

CONDITIONS: Analgesia, Patient-Controlled
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- sufentanil administration intravenously (Experimental): The dose of sufentanil for patient-controlled analgesia is 3.0μg/Kg dissolving in 100ml 0.9% normal saline (NS).The PCA pump is connected to the hand vein.The parameters were set as background dose 1.5 ml/h, PCA dose 1ml, locking time 15 min.
  Interventions: Drug: intravenous sufentanil
- sufentanil administration subcutaneously (Experimental): The dose of sufentanil for patient-controlled analgesia is 3.0μg/Kg dissolving in 100ml 0.9%NS.The PCA pump is connected to the deltoid subcutaneously.The parameters were set as background dose 1.5 ml/h, PCA dose 1 ml, locking time 15 min.
  Interventions: Drug: subcutaneous sufentanil
- hydromorphone administration intravenously (Experimental): The dose of hydromorphone for patient-controlled analgesia is 0.2mg/Kg dissolving in 100ml 0.9%NS.The PCA pump is connected to the hand vein.The parameters were set as background dose 1.5 ml/h, PCA dose 1 ml, locking time 15 min.
  Interventions: Drug: intravenous hydromorphone
- hydromorphone administration subcutaneously (Experimental): The dose of hydromorphone for patient-controlled analgesia is 0.2mg/Kg dissolving in 100ml 0.9%NS.The PCA pump is connected to the deltoid subcutaneously.The parameters were set as background dose 1.5 ml/h, PCA dose 1 ml, locking time 15 min.
  Interventions: Drug: subcutaneous hydromorphone
- sufentanil and dexmedetomidine intravenously (Experimental): The dose of sufentanil, dexmedetomidine,for patient-controlled analgesia is 3.0μg/Kg, dissolving in 100ml 0.9% normal saline (NS).The PCA pump is connected to the hand vein.The parameters were set as background dose 1.5 ml/h, PCA dose 1ml, locking time 15 min.
  Interventions: Drug: intravenous sufentanil and dexmedetomidine
- sufentanil and dexmedetomidine subcutaneously (Experimental): The dose of sufentanil ,dexmedetomidine ,for patient-controlled analgesia is 3.0μg/Kg dissolving in 100ml 0.9%NS.The PCA pump is connected to the deltoid subcutaneously.The parameters were set as background dose 1.5 ml/h, PCA dose 1 ml, locking time 15 min.
  Interventions: Drug: subcutaneous sufentanil and dexmedetomidine
- hydromorphone and dexmedetomidine intravenously (Experimental): The dose of hydromorphone for patient-controlled analgesia is 0.2mg/Kg ,dexmedetomidine ,for patient-controlled analgesia is 3.0μg/Kg dissolving in 100ml 0.9%NS.The PCA pump is connected to the hand vein.The parameters were set as background dose 1.5ml/h, PCA dose 1ml, locking time 15 min.
  Interventions: Drug: intravenous hydromorphone and dexmedetomidine
- hydromorphone and dexmedetomidine subcutaneously (Experimental): The dose of hydromorphone for patient-controlled analgesia is 0.2mg/Kg ,dexmedetomidine ,for patient-controlled analgesia is 3.0μg/Kg dissolving in 100ml 0.9%NS.The PCA pump is connected to the deltoid subcutaneously.The parameters were set as background dose 1.5ml/h, PCA dose 1 ml, locking time 15 min.
  Interventions: Drug: subcutaneous hydromorphone and dexmedetomidine

INTERVENTIONS:
Drug: intravenous sufentanil — The PCA pumps contain sufentanil . And the pump is connected to participants intravenously .
  Other Names: SI
  Arms: sufentanil administration intravenously
Drug: subcutaneous sufentanil — The PCA pumps contain sufentanil. And the pump is connected to participants subcutaneously.
  Other Names: SS
  Arms: sufentanil administration subcutaneously
Drug: intravenous hydromorphone — The PCA pumps contain hydromorphone. And the pump is connected to participants intravenously .
  Other Names: HI
  Arms: hydromorphone administration intravenously
Drug: subcutaneous hydromorphone — The PCA pumps contain hydromorphone. And the pump is connected to participants subcutaneously.
  Other Names: HS
  Arms: hydromorphone administration subcutaneously
Drug: intravenous sufentanil and dexmedetomidine — The PCA pumps contain sufentanil and dexmedetomidine. And the pump is connected to participants intravenously .
  Other Names: SDI
  Arms: sufentanil and dexmedetomidine intravenously
Drug: subcutaneous sufentanil and dexmedetomidine — The PCA pumps contain sufentanil and dexmedetomidine. And the pump is connected to participants subcutaneously.
  Other Names: SDS
  Arms: sufentanil and dexmedetomidine subcutaneously
Drug: intravenous hydromorphone and dexmedetomidine — The PCA pumps contain hydromorphone and dexmedetomidine. And the pump is connected to participants intravenously.
  Other Names: HDI
  Arms: hydromorphone and dexmedetomidine intravenously
Drug: subcutaneous hydromorphone and dexmedetomidine — The PCA pumps contain hydromorphone and dexmedetomidine. And the pump is connected to participants subcutaneously
  Other Names: HDS
  Arms: hydromorphone and dexmedetomidine subcutaneously

SUMMARY:
To explore the effect of different drugs and infusion ways on degree of postoperative comfort.Patients undergoing spinal neoplasm surgery receive different patient controlled analgesia(PCA) drugs postoperatively,one group is sufentanil,the other is hydromorphone. Then each drug group will be divided into two subgroups according to the infusion way,intravenously,subcutaneously. During the patient controlled analgesia period, patients' degree of comfort,pain score,sleep quality, the degree of side reaction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II .

Exclusion Criteria:

* history of severe heart, hepatic or renal disease,
* history of chronic pain condition or opioid use,
* body mass index (BMI) ≤18 or ≥30 kg/m2,
* alcohol or drug abuse,
* relevant drug allergy,
* inability to properly describe postoperative pain,
* inability to use PCA pump.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale of Comfort level | 48 hours after the use of PCA.
  The participants' comfort level of the PCA."0" means extremely comfort, "10" means extremely discomfort.

SECONDARY OUTCOMES:
Ramsay sedation score | 6hours,12hours,24hours and 48 hours after the use of PCA.
  To evaluate the degree of sedation.
The degree of nausea | 6hours,12hours,24hours and 48 hours after the use of PCA.
  "0" means no nausea and vomiting,"1" means only nausea,"2"means nausea and vomiting .
The degree of dizziness | 6hours,12hours,24hours and 48 hours after the use of PCA.
  "0" means no dizziness,"1" means the time of dizziness less than 2 hours,"2" means the time of dizziness more than 2 hours.
Pupil diameter | 6hours,12hours,24hours and 48 hours after the use of PCA.
  The average diameter of both pupils measuring by pupil pen.

OTHER OUTCOMES:
Pittsburgh sleep quality index | 1 day before the surgery,1 month after the surgery.
  The quality of sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hosipital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Wang J, Cui L, Fan L, Wang J. Clinical Effect of Different Drugs and Infusion Techniques for Patient-controlled Analgesia After Spinal Tumor Surgery: A Prospective, Randomized, Controlled Clinical Trial. Clin Ther. 2021 Jun;43(6):1020-1028. doi: 10.1016/j.clinthera.2021.03.019. Epub 2021 May 2. PMID 33952398